CLINICAL TRIAL: NCT06818240
Title: Transcranial Direct Current Stimulation of the Dorsolateral Prefrontal Cortex Enhances Dual-task Performance in People With Stroke
Brief Title: Transcranial Direct Current Stimulation Enhances Dual-task Performance in Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Shamay Ng, Prof., The Hong Kong Polytechnic University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2025_DUAL_STROKE
Record Dates: First submitted 2025-01-23; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Chronic Stroke
Keywords: transcranial direct current stimulation; stroke; dual task
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A constant current of 2 mA was applied for 30 minutes (Active Comparator): In the active tDCS session, a constant current of 2 mA was applied for 30 minutes, with a 30-second ramp-up and ramp-down for comfort.
  Interventions: Device: Active transcranial direct current stimulation
- no active current was applied throughout the stimulation phase (Sham Comparator): For the sham condition, no active current was applied throughout the stimulation phase, except for an electrical current of 1 mA, which was delivered for the first and last 60 seconds, with similar ramping to control for potential sensation bias.
  Interventions: Device: Sham transcranial direct current stimulation

INTERVENTIONS:
Device: Active transcranial direct current stimulation — In the active tDCS session, real stimulation was delivered via a current stimulator (DC-STIMULATOR MC, NeuroConn, Germany) using saline-soaked 4×6 cm² electrodes. The anode was positioned over the left-DLPFC identified as F3 according to the 10-20 international EEG system, and the cathode over the right supraorbital ridge.
  Arms: A constant current of 2 mA was applied for 30 minutes
Device: Sham transcranial direct current stimulation — In the Sham tDCS session, Sham stimulation was delivered via a current stimulator (DC-STIMULATOR MC, NeuroConn, Germany) using saline-soaked 4×6 cm² electrodes. The anode was positioned over the left-DLPFC identified as F3 according to the 10-20 international EEG system, and the cathode over the right supraorbital ridge.
  Arms: no active current was applied throughout the stimulation phase

SUMMARY:
Stroke often impairs lower limb control, resulting in gait abnormalities and difficulties in dual-task performance, such as walking while engaging in cognitive activities. This study examines the effects of a single session of transcranial direct current stimulation (tDCS) targeting the left dorsolateral prefrontal cortex (DLPFC) on dual-task walking performance in individuals with chronic stroke. Using a cross-over design, participants will undergo two sessions (active or sham tDCS, 7 ± 2 days apart) of stimulation at 2 mA for 30 minutes. Walking performance will be measured using single and dual-task conditions combining motor (e.g., 20 m walk) and cognitive tasks (e.g., word association, random number recall). Primary outcomes include walking speed (m/s), stride length (m), and dual-task cost (DTC) for mobility and cognitive speed.

The study aims to evaluate tDCS as a potential tool to reduce DTC, improve dual-task performance, and improve daily function and quality of life in stroke survivors. Results may guide the development of tailored dual-task interventions in stroke rehabilitation.

DETAILED DESCRIPTION:
Stroke often results in impaired control of lower limb movement, leading to abnormal gait patterns. During daily activities, walking in the community typically involves performing additional cognitive tasks simultaneously, such as remembering directions or engaging in social interactions. Individuals with stroke are particularly susceptible to dual-task interference and demonstrate a slower gait speed, decreased walking adaptability (e.g., obstacle avoidance), and poorer cognitive task performance during dual-task walking, which can increase the dual-task cost (DTC). Transcranial Direct Current Stimulation (tDCS) is a potential tool to reduce DTC, leading to behavioral modifications and improved cognitive functions. This study aims to investigate the effects of a single session of tDCS targeting the left dorsolateral prefrontal cortex (DLPFC) on dual-task walking performance in individuals with chronic stroke.

The study will be a repeated measure designed with two testing sessions (same time in a day, 7 ± 2 days apart between sessions). People with stroke fulfilling the inclusion and exclusion criteria will be recruited from the local community. In each session, active or shame tDCS will be administered first, followed immediately by randomly assigned single and dual tasks. The stimulation will be delivered using a current stimulator (DC-STIMULATOR MOBILE, NeuroConn, Germany). The intensity is set at 2 mA for 30 min. The anode will be placed over the left DLPFC (F3 according to the EEG 10/20 system), while the cathode over the contralateral supraorbital ridge. The gait measurement is recorded by the Opal IMU sensor module and MobilityLab system (APDM Inc., USA).

Measurements of mobility will consist of two walking conditions: single-task and dual-task walking. For the walking test, we perform 'Stand and Walk for a 20-meter Round Trip (10 meters each way)(SWR), which consists of standing for 10 s, walking 10 m, turning, and walking 10 m back. The total time (TT) taken to complete one SWR test will be recorded. For the single cognitive tasks, participants will remain seated and perform the following: Random number, Word association, Counting forward, Serial subtraction. The time taken to complete each task will be equivalent to the TT recorded during the SSWR test. Additionally, the number of correct responses and errors made during the cognitive tasks will be recorded for further analysis. For the dual tasks, we will combine motor and cognitive tasks to assess dual-task performance. The specific dual tasks include SWR + Random Number, SWR + Word Association, SWR + Counting Forward, SWR + Serial Subtraction, SWR + Head Turns, and SWR+ Visual Fixation. The time taken to complete each task and the number of correct responses and errors made will be recorded for further analysis.

The primary outcomes include gait speed (m/s), stride length (m), and dual-task costs (DTC) for mobility and cognition speed. Each session will last approximately 60 min, including both tDCS and MobilityLab setup, and rest.

The findings may provide valuable insights into the use of tDCS as an adjunctive treatment for stroke patients. By enhancing the cortical activity of the left DLPFC through tDCS, it is anticipated that the dual-task cost would be reduced, which results in better dual-task performance and an improvement in daily function and overall quality of life for stroke survivors.

ELIGIBILITY:
Inclusion Criteria:

* age between 50 and 80 years
* at least 6 months post-first-ever stroke with unilateral motor deficits
* ability to walk independently for at least 10 m without the use of walking aids
* a score of 24 or higher on the Mini-Mental State Examination (MMSE)

Exclusion Criteria:

* unstable medical conditions, such as heart failure, uncontrolled hypertension, or cancer
* presence of other comorbidities that could interfere with gait
* history of contraindications to tDCS, such as epilepsy or metal implants
* history of head injury, head surgery, or lower limb orthopedic issues

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Gait speed | Immediately after the active/sham tDCS intervention
  Kinematic data will be collected using a motion tracking system, the MobilityLab system (APDM Inc., Portland, OR, USA), and the Opal IMU sensor module (with 128 Hz sampling frequency). A total of eight sensors will be attached with Velcro straps to the sternum of the upper body, the lumbar region, and pairs of thighs, lower legs, and feet. The walking speed (m/s) will be recorded during each walking task.
Stride length | Immediately after the active/sham tDCS intervention
  Kinematic data will be collected using a motion tracking system, the MobilityLab system (APDM Inc., Portland, OR, USA), and the Opal IMU sensor module (with 128 Hz sampling frequency). A total of eight sensors will be affixed using velcro belts, positioned on the sternum of the upper body, at the lumbar region, and on pairs of upper legs, lower legs, and feet. Stride length (m) will be recorded during each walking task.
Cognitive response rate | Immediately after the active/sham tDCS intervention
  Cognitive performance will be evaluated during each task by the number of correct words per second, defined as the response rate (correct responses/second).
DTC- Mobility speed | Immediately after the active/sham tDCS intervention
  The impact of dual-tasking will be quantified by calculating the dual-task cost (DTC) using the following formula: DTC (%) = (dual task outcome measure-single task outcome measure)/single task outcome measure × 100. DTC-mobility speed indicates the variation in speed used under dual-task versus single-task conditions.
DTC- Cognitive speed | Immediately after the active/sham tDCS intervention
  The impact of dual-tasking will be quantified by calculating the dual-task cost (DTC) using the following formula: DTC (%) = (dual task outcome measure-single task outcome measure)/single task outcome measure × 100. For example, DTC-time reflects the variation in time taken to complete the SWR test under dual-task versus single-task conditions. DTC- Cognitive speed represents the variation in response rate under both conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Shamay SM NG, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, China, Hong Kong

IPD SHARING:
Plan to Share IPD: No